CLINICAL TRIAL: NCT02119598
Title: Technical and Clinical Feasibility of Third Generation In-ambulance Telemedicine: Feasibility of AmbulanCe-based Telemedicine (FACT) Study
Brief Title: Feasibility of AmbulanCe-based Telemedicine (FACT) Study
Acronym: FACT
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Raf Brouns, MD, PhD, M.D., Ph.D., Universitair Ziekenhuis Brussel
Other Study IDs: B.U.N. 143201317990
Record Dates: First submitted 2014-04-12; First posted 2014-04-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Acute Stroke
Keywords: Prehospital care; Telemedicine; Ambulance-based telemedicine
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Research on prehospital telestroke systems is recommended by the American Stroke Association, as it may facilitate early stroke diagnosis, assessment of stroke severity and selection of patients for specific stroke treatments

The experience with prehospital telemedicine for assessment of stroke severity is limited. Prehospital telestroke is a very promising concept, facilitating specialized stroke care in very early stage based on integration of bidirectional audiovisual communication with point of care laboratory analysis, vitals and decision support software.

The aim of this prospective study is to investigate the safety, the technical feasibility and the reliability of in-ambulance telemedicine using a prototype third generation telemedicine system (PreSSUB 3.0).

DETAILED DESCRIPTION:
Timely treatment can effectively reduce the burden of stroke and should begin with optimal prehospital stroke care. The slogans 'Time is brain' and 'Competence is brain' adequately point out that acute stroke is a time-critical medical emergency requiring specialized treatment.

Pursuant to ongoing technological developments and in line with the American Stroke Association and the European Stroke Organisation guidelines, the implementation of telestroke for optimizing inhospital stroke care is currently applied in several countries. Research on prehospital telestroke systems is recommended by the American Stroke Association, as it may facilitate early stroke diagnosis, assessment of stroke severity and selection of patients for specific stroke treatments.

The experience with prehospital telemedicine for assessment of stroke severity, however, is limited to the TeleBAT project and two recent pilot studies conducted in healthy volunteers. Prehospital telestroke is a very promising concept, facilitating specialized stroke care in very early stage based on integration of bidirectional audiovisual communication with point of care laboratory analysis, vitals and decision support software.

As part of the Prehospital Stroke Study at the Universitair ziekenhuis Brussel (PreSSUB), we have developed and tested several prototypes for prehospital telemedicine. The current system consists of commercially available hardware and a Web-based telemedicine platform. The data are transmitted to a multimedia server unit over a mobile (ultra)broadband connection (3G or 4G). Data privacy is secured by password-protected logins, role-based access control, and hypertext transfer protocol secure encryption.

The results of a feasibility study using the 4G network in healthy volunteers have recently been reported and feasibility data using the 3G network in healthy volunteers are available.

Building further on the reassuring safety and feasibility data specified above, the next logical step is to evaluate this system for prehospital telemedicine in the real-life situation involving transportation of patients in the Paramedic Ambulance team (PIT)-ambulance to the UZ Brussel.

ELIGIBILITY:
Inclusion Criteria:

* Any patient older than 18 years of age requesting ambulance-based emergency care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient older than 18 years requesting ambulance-based emergency care.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of succesfully executed prehospital teleconsultations | Up to 26 weeks
  A successful prehospital teleconsultation is defined as a personal interaction between a patient in a moving ambulance and a remote teleconsultant, based on wireless audiovisual communication and optional reporting of vital parameters (e.g. blood pressure, blood oxygen saturation, heart rate, glycemia), neurological deficit, key history taking, medication anamnesis, and/or patient identification.

CONTACTS AND LOCATIONS:
Overall Officials: Raf Brouns, M.D., Ph.D., Principal Investigator — Department of Neurology, Universitair Ziekenhuis Brussel, Belgium
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium